CLINICAL TRIAL: NCT07045935
Title: Metabolic Outcomes in Patients With Prolactinomas Under Dopamine Agonist Treatment - A Randomized, Single-Blind Active- Controlled Trial
Brief Title: Metabolic Outcomes in Patients With Prolactinomas Under Dopamine Agonist Treatment
Acronym: ProBOLIC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-00829; kt25Atila
Record Dates: First submitted 2025-06-12; First posted 2025-07-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Prolactinoma
Keywords: hyperprolactinemia; cabergoline; prolactin level; Dopamine agonist; glucose level; Oral Glucose Tolerance Test; hypoprolactinemia
MeSH Terms: conditions — Prolactinoma; Hyperprolactinemia; Prolactin Deficiency, Isolated | interventions — Cabergoline; Dopamine Agonists

STUDY DESIGN:
Intervention Model Description: Randomized, Single-Blind Active-Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors (e.g., study nurses and study physicians) will all remain blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention arm (Cabergoline) (Active Comparator): The experimental intervention arm aims to treat patients (with hyperprolactinemia) with Cabergoline (Dopamine Agonist) by targeting the suppression of prolactin levels (below the normal plasma prolactin range).
  Interventions: Drug: Cabergoline (Dopamine Agonist)
- Control intervention arm (Cabergoline) (Active Comparator): The control intervention arm aims to treat patients (with hyperprolactinemia ) with Cabergoline (Dopamine Agonist) by targeting the normalisation of prolactin levels (within the normal plasma prolactin range).
  Interventions: Drug: Cabergoline (Dopamine Agonist)

INTERVENTIONS:
Drug: Cabergoline (Dopamine Agonist) — Cabergoline is available in tablet form, with doses of 0.5 mg per tablet. The standard dosing for hyperprolactinemia typically starts at 0.25 mg to 0.5 mg per week, which can be gradually increased based on the patient's response, with a usual range of 0.25 mg to 2 mg per week. The dose required to achieve the target prolactin levels (pre- defined for each intervention arm) may vary between patients, so a fixed dose is not specified. This allows for individualized treatment based on each patient's response.

SUMMARY:
This randomized, active-controlled, parallel-arm, single-blind trial is to compare the effects of Dopamine agonists (DA) therapy targeting different established treatment strategies on glucose metabolism assessed by an oral glucose tolerance test.

DETAILED DESCRIPTION:
Prolactinomas are the most common pituitary tumors, leading to hyperprolactinemia, which causes hypogonadism, infertility, and is associated with adverse metabolic effects such as insulin resistance, dyslipidemia, and obesity. Dopamine agonists (DAs), especially cabergoline, are the first-line treatment. They reduce prolactin levels and tumor size effectively. Despite their widespread use, there are no evidence-based guidelines regarding target prolactin levels during DA therapy. Limited evidence suggests that different prolactin levels may have different effects on metabolic health. This trial aims to assess glucose tolerance, insulin sensitivity, and beta-cell function-using OGTT with insulin levels-after 12 months of DA treatment, to target treatment options.

In Switzerland, cabergoline is the preferred DAs for treating hyperprolactinemia.

Cabergoline is available in tablet form, with doses of 0.5 mg per tablet. The standard dosing for hyperprolactinemia typically starts at 0.25 mg to 0.5 mg per week, which can be gradually increased based on the patient's response, with a usual range of 0.25 mg to 2 mg per week.

ELIGIBILITY:
Inclusion Criteria (treatment-naïve patients):

* Diagnosed adult patients (at least 18 years of age) with prolactinoma-induced hyperprolactinemia, defined as a prolactin level ≥ two times the local laboratory maximum and radiographic criteria, based on current guidelines.

Inclusion Criteria (treatment-naïve patients):

* Diagnosed adult patients (at least 18 years of age) with prolactinoma-induced hyperprolactinaemia based on current guidelines.
* Patients treated with cabergoline as DA therapy and prolactin levels within the normal range

Exclusion Criteria:

* alternative explanation for hyperprolactinaemia
* Active substance use disorder within the last six months
* Current or previous psychotic disorder
* Pregnancy or breastfeeding within the last 8 weeks
* Severe hepatic insufficiency or cholestasis

  * Child Pugh C or
  * AST/ ALT > 3 x the upper limit of normal ULN or
  * Cholestasis (total bilirubin > 2x ULN)
* Severe renal impairment (eGFR < 30 ml/min)
* History of pulmonary, pericardial, and/or retroperitoneal fibrotic disorders
* Concomitant treatment with strong or moderate CYP3A4 inhibitors
* Local complications on morphological imaging, related to signs or clinical symptoms which make surgical intervention necessary or a clear patient's preference for surgical treatment
* Gastrointestinal disease or previous surgery: chronic active inflammatory bowel disease, active gastrointestinal ulcer disease, or surgery on the gastrointestinal tract (e.g. sleeve stomach, gastric band)
* Patient incapable of giving informed consent due to cognitive impairment or other reasons (e.g., legal incapacity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
2-hour post-oral glucose tolerance test (OGTT) plasma glucose levels | assessed at 12 months after randomisation
  The OGTT is a test used to assess the ability to process glucose. It involves fasting overnight and then drinking a solution containing a measured amount of glucose (75g). Blood Samples are taken at 120 min after glucose intake.

SECONDARY OUTCOMES:
Change in Insulin sensitivity by MATSUDA Index | measured at time points (0, 30, 60, 90, and 120 minutes) during the OGTT
  The Matsuda Index is a measure used to assess insulin sensitivity from the data obtained during an OGTT. The Index is derived from OGTT data and reflects whole-body insulin sensitivity by incorporating both fasting and postprandial glucose and insulin levels. The formula uses (1) fasting glucose and insulin before the glucose load and (2) mean glucose and mean insulin.
Change in Insulin Sensitivity Index (ISI) | measured at time points (0, 30, 60, 90, and 120 minutes) during the OGTT
  ISI is an OGTT-based measure that quantifies insulin sensitivity using fasting and post-load insulin and glucose values. It is similar to the Matsuda Index but has variations depending on specific formulas. Higher ISI values reflect better insulin action.
Change in Quantitative Insulin Sensitivity Check Index (QUICKI) | measured at time points Screening, Month 6, Month 12, Month 24
  QUICKI is a simple, fasting- based index to estimate insulin sensitivity, calculated as 1 / (log(Fasting Insulin) + log(Fasting Glucose)). Higher values indicate greater insulin sensitivity.
Change in Glycated Haemoglobin (HbA1c) | measured at time points Screening, Month 3, Month 6, Month 12
  HbA1c reflects average blood glucose levels over the past 2-3 months by measuring glucose-bound haemoglobin. It is used for diagnosing and monitoring diabetes, with values ≥6.5% indicating diabetes.
Change in Fasting glucose (mmol/L) | measured at time points Screening, Month 3, Month 6, Month 12
  Fasting glucose measures baseline blood sugar levels after at least 8 hours of fasting. It is a primary diagnostic criterion for diabetes, with ≥7.0 mmol/L indicating diabetes.
Change in Fasting insulin (µU/mL) | measured at time points Screening, Month 3, Month 6, Month 12
  Fasting insulin provides insight into pancreatic insulin secretion and insulin resistance. Elevated levels often indicate insulin resistance, while low levels may suggest beta-cell dysfunction.
Change in C-peptide (nmol/l) | measured at time points Screening, Month 3, Month 6, Month 12
  C-peptide is released in equal amounts to insulin and is used to assess endogenous insulin production
Change in Disposition Index (DI) | measured at time points Screening, Month 3, Month 6, Month 12
  The DI integrates beta-cell function and insulin sensitivity, calculated as insulin secretion × insulin sensitivity. It reflects how well beta-cells compensate for insulin resistance, with lower values indicating a higher risk of diabetes.
Change in plasma prolactin levels (ng/mL) | measured at time points Screening, Month 3, Month 6, Month 12
  Change in plasma prolactin levels (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Atila, Dr., Principal Investigator — University Hospital Basel, Dept. of Endocrinology, Metabolism & Diabetes
Locations (1):
- University Hospital Basel, Dept. of Endocrinology, Metabolism & Diabetes, Basel, Switzerland